CLINICAL TRIAL: NCT03899961
Title: The Clinical Carbetocin Myocardium Trial Part 2
Brief Title: Carbetocin Myocardium Trial 2014 Part 2
Acronym: CMT2014/2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Leiv Arne Rosseland, Professor PhD MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014/1210
Record Dates: First submitted 2019-01-30; First posted 2019-04-02 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Complications
Keywords: cesarean delivery; blood loss; troponin
MeSH Terms: conditions — Pregnancy Complications; Hemorrhage | interventions — Oxytocin; carbetocin

STUDY DESIGN:
Intervention Model Description: The study is a parallel, randomized, blinded phase 4 study (safety)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Active Comparator): Oxytocin 2.5 U i.v.
  Interventions: Drug: Oxytocin
- Carbetocin (Experimental): Carbetocin 100 µg i.v.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 2.5 U i.v.
  Arms: Oxytocin
Drug: Carbetocin — Carbetocin 100 µg i.v.
  Arms: Carbetocin

SUMMARY:
Carbetocin has been in clinical use in EU for some years and the efficacy is documented in several RCTs. Circulatory adverse events leading to death has been reported after intravenous injection of oxytocin. Some studies indicate that oxytocin may lead to dose dependent ischemic ECG changes, prolongation of QT time and liberation of biomarkers of myocardial cell death. Previously the investigators have demonstrated comparable vasodilatory effects of oxytocin and carbetocin. There is no clinical study comparing the specific myocardial effects of oxytocin with carbetocin. It may have great impact on the choice of standard medication if the cardiotoxicity of carbetocin is lower compared with oxytocin. The study of potential cardiotoxicity has to be performed in healthy women. Knowing that millions of laboring women have had uneventful injections of oxytocin and carbetocin after delivery, there is probably no reason to fear long lasting negative effects of either drug. If there are differences in cardiotoxicity, this new information should be taken into consideration when planning delivery in pregnant women with heart disease.

DETAILED DESCRIPTION:
Background -Treatment Caesarean delivery is a commonly performed surgical procedure. Uterus contraction after delivery of the baby is necessary to avoid excessive bleeding.

Background - Therapeutic Information Adequate uterus contraction after delivery of the baby is necessary to avoid excessive bleeding. Prophylactic administration of an oxytocin receptor agonist is first line practice. Intravenous injection of oxytocin has been the standard procedure but serious cardiovascular adverse events have been reported. Lowering the dose or administering the drug as a 5 minute infusion may increase safety. Carbetocin, a synthetic oxytocin receptor agonist, has significantly longer half life and may reduce blood loss compared with oxytocin. The hemodynamic vasodilatory effects are comparable to oxytocin, but potential differences in adverse effects on myocardium are not well described yet.

Pre-Clinical & Clinical Experience with Carbetocin (IMP) and Oxytocin Carbetocin has been in clinical use in EU for some years and the efficacy is documented in several RCTs. In the proposed study, carbetocin will be used within the conditions of the marketing authorization. Oxytocin is the first line treatment and prophylaxis in Norway and most countries in the world. According to recently published guidelines from EU drug authorities (EMA), oxytocin should be given as a slow, 5-minute infusion in order to avoid hypotension. This has so far not been implemented in Norway. The pre-clinical and clinical experience of the two drugs are summarized in the Summaries of Product Characteristics.

Rationale for the Study Pregnancy and delivery is a natural process, but for many women this period is stressful and not without risks of morbidity, and even mortality. Circulatory adverse events leading to death has been reported after intravenous injection of oxytocin. Some studies indicate that oxytocin may lead to dose dependent ischemic ECG changes, prolongation of QT time and liberation of biomarkers of myocardial cell death. Previously the investigators have demonstrated comparable vasodilatory effects of oxytocin and carbetocin. There is no clinical study comparing the specific myocardial effects of oxytocin with carbetocin. It may have great impact on the choice of standard medication if the cardiotoxicity of carbetocin is lower compared with oxytocin. The study of potential cardiotoxicity has to be performed in healthy women. Knowing that millions of laboring women have had uneventful injections of oxytocin and carbetocin after delivery, there is probably no reason to fear long lasting negative effects of either drug. If there are differences in cardiotoxicity, this new information should be taken into consideration when planning delivery in pregnant women with heart disease.

STUDY OBJECTIVES The aims of this study are to compare 0h (before C-section) plasma concentrations of Troponin I (high sensitive methods) with a second measurement of plasma concentration of Troponin I drawn within an interval of 6 to 10 hours after administration of study drug, in elective healthy C-section patients randomized to oxytocin 2.5 U or carbetocin 100 µg, 1 minute injection immediately after delivery.

Primary Endpoint Primary outcome measure is the difference in plasma concentration of Troponin I from baseline (0h) to the second measurement 6-10 hours after test drug administration, according to treatment allocation. Plasma concentrations will be collected before C-section, and at an interval of 6-10 h after test drug administration.

Secondary Endpoints

* Other myocardial biomarkers
* Uterus tone evaluated repeatedly
* Blood loss (estimated calculated blood loss)
* Postoperative pain and side effects.
* BP, heart rate and ECG changes

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant women age 18 to 50
2. Singleton pregnancy at gestational age 36 weeks or more
3. Able to read and understand Norwegian.
4. Patients will be recruited from the general population at the birth clinic at Oslo University Hospital or the birth clinic of Akershus University Hospital. Signed informed consent form (ICF) and expected cooperation of the patients for the treatment and follow up will be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

1. Patients with placenta pathology such as praevia, accreta, pre-eclampsia
2. Patients with bleeding disorders including vonWillebrand disease type I.
3. Known intolerance to one of the two drugs.
4. Patients with prolonged QT-time or other serious cardiac diseases.
5. Liver or kidney failure.
6. Epilepsy.
7. Any medical reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Sem-Thagaard, MD, Study Director — Oslo Universitetssykehus
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog
  - Division of Anaesthesia and Intensive Care Medicine, Oslo University Hospital - Rikshospitalet, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bekkenes ME, Jorgensen MM, Jacobsen AF, Fagerland MW, Rakstad-Larsen H, Aaberge L, Klingenberg O, Steinsvik T, Asphaug L, Rosseland LA. Effects of Prophylactic Oxytocin or Carbetocin on Troponin Release and Postpartum Haemorrhage at Planned Caesarean Delivery: A Double-Blind Randomised Controlled Trial. BJOG. 2025 Nov;132(12):1742-1752. doi: 10.1111/1471-0528.18312. Epub 2025 Aug 7. PMID 40772429
- [Derived] Bekkenes M, Jorgensen MM, Flem Jacobsen A, Wang Fagerland M, Rakstad-Larsen H, Solberg OG, Aaberge L, Klingenberg O, Steinsvik T, Rosseland LA. A study protocol for the cardiac effects of a single dose of either oxytocin 2.5 IU or carbetocin 100 microg after caesarean delivery: a prospective randomized controlled multi-centre trial in Norway. F1000Res. 2021 Sep 27;10:973. doi: 10.12688/f1000research.73112.2. eCollection 2021. PMID 34745566

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Carbetocin
Started | 121 | 119
Completed | 112 | 103
Not Completed | 9 | 16
Not completed — -delivery prior to | 2 | 7
Not completed — req general anesth | 1 | 2
Not completed — capacity | 5 | 6
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Modified ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Carbetocin | Total
Number analyzed (Participants) | 112 | 103 | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 103 | 215
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 34.5 [23.4 to 50.9] | 35.0 [24.1 to 47.5] | 34.8 [23.4 to 50.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 103 | 215
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 112 | 103 | 215
Region of Enrollment [Count of Participants; unit: Participants]
  Norway | 112 | 103 | 215
Troponin I [Median (Full Range); unit: ng/L] | 1.0 [1.0 to 48.7] | 1.0 [1.0 to 19.2] | 1.0 [1.0 to 48.7]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration Troponin I
Description: Group difference in plasma concentration of Troponin I
Time Frame: 8 hours
Population: Biobank sample
Measure: Median (Full Range); unit: ng/L
Arm/Group | Oxytocin | Carbetocin
Number analyzed (Participants) | 109 | 99
ng/L | 1.2 [1.0 to 47.0] | 1.2 [1.0 to 19.5]
Statistical Analysis 1: Comparison: Oxytocin vs Carbetocin; Median regression model for the change from baseline, model was adjusted for treatment, bootstrap was used for the confidence interval; Test type: Superiority — Median regression model for the change from baseline, model was adjusted for treatment, bootstrap was used for the confidence interval; p = 0.05, Median regression model for the change f — Median regression model for the change from baseline, model was adjusted for treatment, bootstrap was used for the confidence interval; Median Difference (Net) = 0, 95% CI 2-sided [-1.09 to 1.09]

2. Secondary Outcome: Blood Loss
Description: Blood loss estimated by hemoglobin
Time Frame: 10 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Oxytocin | Carbetocin
Number analyzed (Participants) | 112 | 103
mL | 386 (369) | 361 (435)

3. Secondary Outcome: Uterine Tone Grade
Description: Peroperative assessment of uterine tone grade 0-10 where 0 is no tonus, 10 is maximal tonus
Time Frame: 5 min
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Oxytocin | Carbetocin
Number analyzed (Participants) | 112 | 103
score on a scale | 7 [4 to 10] | 8 [4 to 10]

4. Secondary Outcome: Side Effects
Description: Perioperative side effects, such as palpitations
Time Frame: 10 min
Population: Side effects in the time period 5 to 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Carbetocin
Number analyzed (Participants) | 112 | 103
Participants | 50 | 55

ADVERSE EVENTS:
Time Frame: 48 h
Description: MedDRA v4
Arm/Group | Oxytocin | Carbetocin
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/103
Other Adverse Events (participants affected / at risk) | 50/112 | 55/103
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=112) | Carbetocin (N=103)
Feeling hot (General disorders) | 23 (23) | 27 (27) — Feeling of warmth
Chest pain (Cardiac disorders) | 12 (12) | 4 (4)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (9)
palpitations (Cardiac disorders) | 7 (7) | 3 (3)
flushing (Vascular disorders) | 11 (11) | 8 (8)
headache (Nervous system disorders) | 6 (6) | 8 (8)
dry mouth (Gastrointestinal disorders) | 1 (1) | 14 (14)
nausea (Gastrointestinal disorders) | 8 (8) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT03899961/Prot_005.pdf
  • Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT03899961/SAP_006.pdf